CLINICAL TRIAL: NCT04477538
Title: The Impact of Operative Approach on Long Term Function Outcomes and Pain in Implant-based Post-mastectomy Breast Reconstruction
Brief Title: Long Term Function Outcomes and Pain in Implant-based Post-mastectomy Breast Reconstruction
Status: Terminated | Type: Observational
Why Stopped: PI decision
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202006199
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Post-mastectomy Breast Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with prepectoral reconstruction: -Participants will complete the post-mastectomy breast reconstruction physical well-being survey
  Interventions: Other: Post-mastectomy breast reconstruction physical well-being survey
- Participants with postpectoral reconstruction: -Participants will complete the post-mastectomy breast reconstruction physical well-being survey
  Interventions: Other: Post-mastectomy breast reconstruction physical well-being survey

INTERVENTIONS:
Other: Post-mastectomy breast reconstruction physical well-being survey — -The survey will ascertain: function status (BREAST Q - Physical Well Being Module and PROMIS upper extremity function), former interaction with physical or occupational therapy, amount of narcotics taken weekly due to chest/neck/breast pain, amount of Tylenol or similar anti-inflammatories taken weekly due to chest/neck/breast pain, and amount of muscle relaxants taken weekly due to chest/neck/breast pain.

SUMMARY:
The objective of this proposal is to broadly assess patient physical functioning following breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 18 years of age
* Had a mastectomy for breast cancer or cancer prevention any time between 01/01/2010 and 06/30/2021.
* Has undergone breast reconstruction surgery with plastic surgery faculty at the Washington University School of Medicine Division of Plastic and Reconstructive Surgery.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

-Known distant metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who undergone breast reconstruction surgery with plastic surgery faculty at the Washington University School of Medicine Division of Plastic and Reconstructive Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Compare the physical well-being Q-score derived from the BREAST-Q between the two groups | Completion of study (estimated to be 30 months)
  The physical well-being module is one of the domains of the BREAST-Q that can be administered in isolation. Patients answer specific questions with answers that range from 1-4 to 1-5. Upon completion of this component of the survey, a physical well-being-specific numerical score is generated. This is then converted, based on previously published Rasch-modeling to generate a Q-score whose values range from 0-100. This same approach is used for all other domains of the BREAST-Q. Pre- versus postoperative Q-scores for physical well-being can be directly compared to study the impact of surgery on physical well-being. Similarly, the physical-well-being domain can be readministered to provide a longitudinal assessment of physical function over time.

SECONDARY OUTCOMES:
Satisfaction with outcome | Completion of study (estimated to be 30 months)
  -The satisfaction with outcome module is one of the domains of the BREAST-Q. Patients answer specific questions with answers that range from 1-3. Upon completion of this component of the survey, a specific numerical score is generated. This is then converted, based on previously published Rasch-modeling to generate a Q-score whose values range from 0-100.
Satisfaction with breasts | Completion of study (estimated to be 30 months)
  -The satisfaction with breast module is one of the domains of the BREAST-Q. Patients answer specific questions with answers that range from 1-4. Upon completion of this component of the survey, a specific numerical score is generated. This is then converted, based on previously published Rasch-modeling to generate a Q-score whose values range from 0-100.
Upper extremity function as measured by PROMIS Upper Extremity Short Form 7a | Completion of study (estimated to be 30 months)
  -Questions regarding upper extremity function as reported by patient. Answers range from 5=without any difficulty to 1=unable to do. The total score ranges from 5-35.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Myckatyn, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu